CLINICAL TRIAL: NCT03464695
Title: Automated Oxygen Delivery by O2matic to Patients Admitted With an Exacerbation in COPD
Acronym: O2MATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Ejvind Frausing Hansen, Chief Physician, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: O2MATIC-COPD
Record Dates: First submitted 2018-03-02; First posted 2018-03-14 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: COPD Exacerbation; Hypoxia; Hyperoxia; Respiratory Failure; Respiratory Insufficiency; Copd Exacerbation Acute
Keywords: closed-loop; oxygen treatment
MeSH Terms: conditions — Hypoxia; Hyperoxia; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O2matic (Active Comparator): Oxygen administered by O2matic. Automatic adjustment based on continuous measurement of SpO2.
  Interventions: Device: O2matic
- Manual (No Intervention): Oxygen administered by manual control based on nurse's intermittent measurement of SpO2.

INTERVENTIONS:
Device: O2matic — Continous measurement of SpO2 during an admission with COPD, and closed-loop control of oxygen-delivery to maintain SpO2 within a target interval.
  Arms: O2matic

SUMMARY:
The aim of the study is to examine if automated oxygen delivery with O2matic is better than manually controlled oxygen therapy for patients admitted to hospital with an exacerbation in Chronic Obstructive Pulmonary Disease (COPD).

O2matic is a closed -loop system based on continuous non-invasive measurement of pulse and oxygen-saturation that is processed in an algorithm that controls the flow of oxygen to the patient.

The primary hypothesis is that O2matic increases time within acceptable oxygen-saturation interval. Secondary hypotheses are that O2matic compared to manual control reduces time with severe hypoxia (SpO2 < 85 %), hypoxi (SpO2 below intended interval) and hyperoxia (SpO2 above intended interval).

DETAILED DESCRIPTION:
Closed-loop control of oxygen therapy is described in the literature used for preterm infants, trauma patients, medical emergency use and patients with COPD. For the latter, closed-loop therapy has been used for patients admitted to hospital with an exacerbation, for domiciliary oxygen use and during exercise. O2matic is a closed-loop system that is based on continuous and non-invasive measurement of pulse, oxygen-saturation and respiratory frequency. The algorithm in O2matic controls oxygen delivery with the aim of keeping the saturation within the desired interval, which could be 88-92 % for COPD-patients in accordance with international guidelines on this topic. Saturation interval can be set for the individual patients, as can the range of acceptable oxygen-flow. If saturation or oxygen-flow can't be maintained within the desired intervals an alarm will sound.

All studies on closed-loop systems have shown that this method is better than manually control by nurse to maintain saturation within the desired interval. Furthermore, some studies have indicated that closed-loop has the possibility to reduce admission time and to reduce time spent with oxygen therapy, due to more efficient and fast withdrawal from oxygen supplementation.

In the present study O2matic will be tested versus manual control, for patients admitted with an exacerbation in COPD, and in need of supplemental oxygen. During the study the patients will either have oxygen controlled with O2matic or manually by nursing staff. All patients will have continuous logging of pulse, oxygen-saturation and oxygen-flow with O2matic, but only in the O2matic active group, the algorithm will control oxygen-delivery.

The primary hypothesis will be tested, which is that O2matic is better than manual control for maintaining oxygen-saturation within the desired interval and reducing time with unintended hypoxia and hyperoxia. For this purpose 20 patients will be included in a crossover design with 4 hours of O2matic-controlled oxygen treatment and 4 hours with manually titrated oxygen with a 16 hours washout between periods.

No safety issues has been reported in the literature. Before use O2matic will be approved by The Danish Medicines Agency, The Ethics Committee in the Capital Region of Denmark and by the regional Data Protection Board. The study will be conducted according to GCP standards with independent monitoring. All adverse events and serious adverse events will be monitored and serious adverse events will be reported to Danish Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

* COPD verified by FEV1/FVC < 0,70
* Admission due to exacerbation in COPD
* COPD exacerbation and pneumonia can be included
* Duration of admission > 48 hours
* Need for oxygen supplementation at inclusion (SpO2 <= 88 % without O2 suppl.)
* Cognitively able to participate in the study
* Willing to participate and give informed consent.

Exclusion Criteria:

* Need or anticipated need for mechanical ventilation (except intermittent CPAP)
* Major co-morbidities (cancer, heart disease, thromboembolic disease, uncontrolled diabetes)
* Asthma or other respiratory condition requiring higher SpO2 than normal for COPD- patients
* Pregnancy
* Acute thromboembolic disease (< 2 weeks)
* Cognitive barriers for participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Time within SpO2-interval | 4 hours
  Fraction of time where SpO2 is kept within desired interval (e.g. 88-92 %) relative to time with SpO2-signal.

SECONDARY OUTCOMES:
Time with severe hypoxia | 4 hours
  Fraction of time where SpO2 is below 85 % relative to time with SpO2 signal
Time with hypoxia | 4 hours
  Fraction of time where SpO2 is below intended interval but not below 85 % relative to time with SpO2 signal
Time with hyperoxia | 4 hours
  Fraction of time where SpO2 is above intended interval relative to time with SpO2 signal

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Vestbo, DMSc, Study Chair — Manchester University Hospital; Ejvind Frausing Hansen, MD, Principal Investigator — Hvidovre University Hospital, Copenhagen
Locations (2):
- Denmark (2):
  - Gentofte University Hospital, Hellerup
  - Hvidovre University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claure N, Bancalari E. Closed-loop control of inspired oxygen in premature infants. Semin Fetal Neonatal Med. 2015 Jun;20(3):198-204. doi: 10.1016/j.siny.2015.02.003. Epub 2015 Mar 12. PMID 25773271
- [Background] Johannigman JA, Branson R, Lecroy D, Beck G. Autonomous control of inspired oxygen concentration during mechanical ventilation of the critically injured trauma patient. J Trauma. 2009 Feb;66(2):386-92. doi: 10.1097/TA.0b013e318197a4bb. PMID 19204511
- [Background] L'Her E, Dias P, Gouillou M, Riou A, Souquiere L, Paleiron N, Archambault P, Bouchard PA, Lellouche F. Automatic versus manual oxygen administration in the emergency department. Eur Respir J. 2017 Jul 20;50(1):1602552. doi: 10.1183/13993003.02552-2016. Print 2017 Jul. PMID 28729473
- [Background] Lellouche F, Bouchard PA, Roberge M, Simard S, L'Her E, Maltais F, Lacasse Y. Automated oxygen titration and weaning with FreeO2 in patients with acute exacerbation of COPD: a pilot randomized trial. Int J Chron Obstruct Pulmon Dis. 2016 Aug 24;11:1983-90. doi: 10.2147/COPD.S112820. eCollection 2016. PMID 27601891
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Background] Rice KL, Schmidt MF, Buan JS, Lebahn F, Schwarzock TK. AccuO2 oximetry-driven oxygen-conserving device versus fixed-dose oxygen devices in stable COPD patients. Respir Care. 2011 Dec;56(12):1901-5. PMID 22288082
- [Result] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955
- See also: Open access to paper with results in Int J Chron Obstruct Pulmon Dis — https://www.dovepress.com/automated-oxygen-control-with-o2maticreg-during-admission-with-exacerb-peer-reviewed-article-COPD